CLINICAL TRIAL: NCT01943513
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Effect of Intravenous BIIB023 (Anti-TWEAK) on Lower Limb Muscle Mass and Strength During and After Knee-Joint Immobilization in Healthy Male Volunteers
Brief Title: A Study of the Effect of BIIB023 on Muscle Atrophy in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 211HV103
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
Keywords: Muscle Disuse Atrophy
MeSH Terms: conditions — Muscular Disorders, Atrophic | interventions — BIIB023; Cytokine TWEAK; Antibodies, Monoclonal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIIB023 (Experimental): Participants receive intravenous (IV) infusions of BIIB023
  Interventions: Biological: BIIB023
- Placebo (Placebo Comparator): Participants receive intravenous (IV) infusions of placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: BIIB023 — Intravenous (IV) infusions
  Other Names: (anti-TWEAK [TNF-related Weak Inducer of Apoptosis] monoclonal antibody)
  Arms: BIIB023
Biological: Placebo — Matched placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine whether muscle atrophy induced by immobilization of the lower limb can be attenuated by BIIB023 in healthy male volunteers. The secondary objectives of this study in this study population are:

* To determine whether muscle weakness induced by immobilization of the lower limb can be attenuated by BIIB023
* To assess the effect of BIIB023 on the recovery of muscle mass and strength after immobilization
* To assess the effect of BIIB023 on histological markers of muscle atrophy and regeneration
* To assess the effect of BIIB023 on muscle bioenergetics based on oxidative metabolism recovery kinetics
* To evaluate the safety and tolerability of BIIB023

ELIGIBILITY:
Key Inclusion Criteria:

* Deemed healthy as determined by the Investigator based on medical history, 12-lead electrocardiogram, vital signs, and clinical laboratory parameters at Screening, and physical examination at Baseline
* Body mass index (BMI) between 18.5 and 32 kg/m2, inclusive, at the time of Screening
* Willing to abstain from using tobacco and tobacco-containing products during the study
* Willing to limit the intake of alcohol to no more than 2 units per day throughout the study; exceptions are 48 hours prior to Screening, 48 hours prior to Day 1, and during the in-clinic immobilization period when no alcohol will be permitted. One unit of alcohol is defined as 12 fluid ounce (fl oz) of beer, 5 fl oz of wine, or 1.5 fl oz of liquor
* Willing to maintain a regular diet for the duration of the study and a recreational level of physical activity defined as participation in an exercise program or other physical activity at a level of intensity that does not exceed the level prior to study entry
* Practice effective contraception during the study and be willing and able to continue contraception for at least 6 months after the last dose of study treatment.

Key Exclusion Criteria:

* History of or positive test result at Screening for human immunodeficiency virus (HIV).
* History or positive test result at Screening for hepatitis C virus (HCV) antibody or hepatitis B virus (defined as positive for hepatitis B surface antigen [HBsAg] or hepatitis B core antibody [HBcAb]).
* History of tuberculosis (TB) or a positive QuantiFERON®-TB Gold test. There must be no other clinical evidence of TB on physical examination of the subject.
* Use of tobacco or tobacco-containing products within 3 months prior to Screening
* Known history of thrombophilia, hypercoagulopathy, or prior history of deep vein thrombosis (DVT) or pulmonary embolism (PE)
* History of physical activity consistent with endurance training or resistance training within 6 months prior to Screening
* Any back, leg, knee, or shoulder complaints that may interfere with the use of crutches
* Prolonged travel (more than 6 hours) within 2 weeks prior to randomization.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Percentage change in the magnitude of muscle atrophy | between Day 14 and Day 42

SECONDARY OUTCOMES:
Percentage change in the magnitude of muscle atrophy, measured by T1W-MRI analysis of the CSA of the triceps surae muscles of the immobilized limb | between Day 14 and Day 42
Percentage change in isometric knee-extension strength (torque), measured by dynamometry | between Day 14 and Day 42
Percentage change in isometric plantar-flexion strength (torque), measured by dynamometry | between Day 14 and Day 42
Percentage change in total CSA of Type I and II fibers, measured by histological analysis of muscle biopsy | between Day 14, Day 21, and Day 42
Change in density of satellite cells and other molecular markers of muscle regeneration, measured by histological analysis of muscle biopsy | between Day 14, Day 21, and Day 42
Change in the recovery of muscle oxidative metabolism, measured by near-infrared spectroscopy (NIRS) of the quadriceps femoris muscles | between Day 14 and Day 42
The number of participants that experience Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 156

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Evansville, Indiana, United States